CLINICAL TRIAL: NCT00399347
Title: Prevalence of Diabetes Mellitus in Ethiopian Community in Israel: an Update
Brief Title: Prevalence of Type 2 Diabetes Mellitus in Ethiopian Community in Israel: an Update
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 4940706
Record Dates: First submitted 2006-11-12; First posted 2006-11-14 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus, prevalence , Ethiopians Jews, Israel
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The prevalence and incidence of diabetes has been reported to vary among populations.Immigrants groups as that have undergone significant life-style changes tend to develop diabetes within a short time. The aim of the study is to assess the prevalence of diabetes mellitus in Ethiopian population ,15-20 years after immigration in Israel.

DETAILED DESCRIPTION:
The study will be conducted in three primary care clinics of the Jezreel Valley (Omer, Givat Hamore and Afula Illit). The computerized medical charts of 500 Ethiopian adults will be reviewed. The following information will be obtained: age, date of arrival in Israel, known history of diabetes, hyperlipidemia, hypertension or other disease, drug therapy, body weight, blood pressure. Following laboratory data will be retrieved: blood glucose, HbA1c, lipid levels , creatinine and uric acid. The criteria used for the definition of diabetes will be based on the criteria proposed by the American Diabetes Association .

ELIGIBILITY:
Inclusion Criteria:

* Male and female Ethiopians Jews who immigrate in Israel in 1991 and were 18 years old or more at immigration.

Exclusion Criteria:

* Type 1 diabetes Mellitus

Min Age: 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of specific region
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2005-01; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ishay MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- Primary care clinics, Afula, Israel